CLINICAL TRIAL: NCT00735098
Title: The Effects of Home-Based Rehabilitation Treatments Among Persons With Symptomatic Knee Osteoarthritis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zululand (Other)
Responsible Party: Principal Investigator, Matthew W. Rogers, MS, Doctoral Student, University of Zululand, University of Zululand
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KneeOAExercise-2
Record Dates: First submitted 2008-08-12; First posted 2008-08-14 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-02

CONDITIONS: Osteoarthritis
Keywords: Knee Osteoarthritis; arthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Arthritis | interventions — Resistance Training; Control Groups

STUDY DESIGN:
Who Masked: Participant

ARMS (4):
- 1 (Experimental): KBA exercise protocol
  Interventions: Other: KBA exercise
- 2 (Experimental): strength training exercise protocol
  Interventions: Other: strength training exercise
- 3 (Experimental): KBA and strength training protocol
  Interventions: Other: KBA and strength training
- 4 (Sham Comparator)
  Interventions: Other: Control group

INTERVENTIONS:
Other: KBA exercise — KBA exercise protocol, 3 times per week for 8 weeks
  Arms: 1
Other: strength training exercise — strength training exercise, 3 times per week for 8 weeks
  Arms: 2
Other: KBA and strength training — KBA and strength training exercise, 3 times per week for 8 weeks
  Arms: 3
Other: Control group — 8 week control group
  Arms: 4

SUMMARY:
Knee Osteoarthritis (OA) is one of the most frequent causes of physical disability and pain among adults. Recent evidence suggests that shorter exercise programs that incorporate kinesthesia, balance and agility (KBA) techniques may result in more rapid symptom relief and functional improvements in comparison to traditional therapeutic exercise. KBA techniques are designed to improve dynamic joint stability by using a series of activities which challenge balance and coordination. To determine the independent effects of KBA training on functional abilities, it is necessary to test it as a training program unto itself. The proposed clinical trial is designed to do this by using three training groups: KBA only; lower extremity strength training only; and a combination of the two. The total exercise time and intensity of each condition will be approximately equal. A non-exercise group will control for any effects related to the testing procedures and the passage of time. Community volunteer men and women age 50 and over with physician diagnosed symptomatic knee OA will participate.

ELIGIBILITY:
Inclusion Criteria:

* Aged 50 years or over of either gender
* Self-reported knee pain
* Physician diagnosed tibiofemoral OA, unilateral or bilateral, per ACR guidelines
* Demonstrated minimal knee OA related dysfunction per WOMAC score
* Not engaged in a regular leg exercise program for minimum of 6 months

Exclusion Criteria:

* High risk health status per (e.g.) ACSM guidelines
* Inability to obtain physician release for exercise
* Unresolved balance disorder
* Unresolved neurological disorder
* History of knee surgery or major knee trauma injury
* Hip or ankle instability, excessive weakness, surgery or major trauma injury
* Hip or knee replacement
* Intra-articular joint injection within 4 weeks of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
(WOMAC) self assessment of physical function | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew W Rogers, MS, Principal Investigator — University of Zululand
Locations (1):
- University of Zululand, St. Petersburg, Florida, United States